CLINICAL TRIAL: NCT05426668
Title: Validation of the TheraSure CNI-Monitor Under Immuno-checkpoint-therapy (Hereinafter: "Immunotherapy") in NSCLC in Palliative Therapy
Acronym: CNI-Monitor
Status: Recruiting | Type: Observational
Sponsor: Karsten Gavenis (Other)
Collaborators: Chronix Biomedical Corporation (Industry)
Responsible Party: Sponsor-Investigator, Karsten Gavenis, on behalf of Principal Investigator Dr. Overbeck, University Medical Center Goettingen
Organization: University Medical Center Goettingen (Other)
Other Study IDs: 2021-01519
Record Dates: First submitted 2022-01-27; First posted 2022-06-22 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
This is a prospective, non-interventional, national study planned at three centers for patients with non-curative NSCLC receiving immunotherapy.

At present, PD-L1 expression or tumor mutation burden serve as surrogate parameters for response to immunotherapy. However, the problem for clinicians is that not all patients with positive findings respond to this form of therapy.

Cell-free DNA (cf-DNA) can be detected in blood plasma. Tumor cells almost always have chromosomal instabilities (or "copy-number variations" (CNV)), which can be detected using next-generation sequencing (NGS), also in the cf-DNA. These CNV can be quantified and given as a cf-DNA copy number instability score (CNI value). TheraSure CNI-Monitor is a highly sensitive method that can detect as little as 0.5% tumor DNA in plasma.

In preliminary work in a cohort of 56 patients with various types of cancer (including: breast, colon, lung, ovary, melanoma) in advanced stages, the TheraSure CNI monitor was already evaluated in the monitoring of immunotherapy. In 51 of the 56 patients, increased CKD values were measured before the start of therapy compared to a normal group of 126 individuals. To predict the success of the therapy, further blood samples were used after the first and second therapy cycle and threshold values were set for the minimal expected decrease in the CNI value in the event of therapy response. A therapy failure could be predicted with a high positive predictive value, cases of hyperprogression could be detected earlier than by routine imaging. In addition, pseudoprogression could be distinguished from true progression using the CNI value.

The CNI monitor on cell-free DNA is to be used prospectively in 170 patients. The primary objective of the study is the prediction of primary progression under immunomonotherapy (defined as PD within 6 months after RECIST) with a predictive value for progression (PPV) of ≥50%.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age ≥18 years
* NSCLC, non-curatively treatable stage III or stage IV with palliative treatment indication
* Immunocheckpoint-therapy for malignant disease (Immunotherapy as monotherapy, double immunotherapy or combination with chemotherapy)

Exclusion Criteria:

* Person is unable to understand the nature, importance and scope of the clinical trial
* Participation in an interventional study
* Hb value <9g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with incurable stage III or stage IV NSCLC on immunotherapy
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
PD | 6 months
  The TheraSure CNI-Monitor predicts primary progression on immunomonotherapy (defined as PD within 6 months acc. to RECIST) with a predictive value for progression (PPV) of ≥50%.

SECONDARY OUTCOMES:
PFS | 6 months
  The TheraSure CNI-Monitor predicts progression-free survival (PFS) in cancer patients receiving immunotherapy. The aim is to determine a significantly different (p<.05) hazard ratio with a describable dichotomized result of the cell-free tumor DNA.
OS | 6 months
  The TheraSure CNI-Monitor predicts overall survival (OS) in cancer patients receiving immunotherapy. The aim is to determine a significantly different (p<.05) hazard ratio with a describable dichotomized result of the cell-free tumor DNA.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - University Medical Center Göttingen, Göttingen, Lower Saxony
  - Medizinische Hochschule Hannover, Hanover
  - Pius-Hospital Oldenburg, Oldenburg